CLINICAL TRIAL: NCT02316288
Title: Preliminary Test of an Integrative Intervention to Alleviate Chronic Pain and Improve Quality of Life
Brief Title: Development of a Couple-based Mindfulness Intervention for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Annmarie Cano, Professor; Associate Chair, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R21AT007939-01A1 (NIH)
Record Dates: First submitted 2014-12-04; First posted 2014-12-12 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapy (Experimental): Mindfulness and Acceptance Therapy
  Interventions: Behavioral: Mindfulness and Acceptance Therapy
- Education (Active Comparator): Health Education
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Mindfulness and Acceptance Therapy — Couples will learn psychological flexibility skills including mindfulness, acceptance, and values-based action as well as relational flexibility skills including empathic listening and responding during weekly 1.5-hour long sessions over the course of this 6-week intervention.
  Arms: Therapy
Behavioral: Health Education — Couples will learn about chronic pain including causes, consequences, and how to talk with their health care professionals about their pain during weekly 1.5-hour long sessions over the course of this 6-week program.
  Arms: Education

SUMMARY:
Chronic pain is a costly public health problem that is associated with poor quality of life. Previous research has demonstrated extensive evidence showing that pain coping is not manifested by patients in isolation but within the context of significant relationships such as marriage. For instance, a partner may avoid or reject their partners' negative emotions about pain, provide unempathic responses to their partners' pain, or change their thoughts about pain. The patient's pain experience and the couples' relationship also have a cyclical relationship, in which both can affect each other and the overall quality of life for both partners. Currently, current clinical practice does not target both partners to alleviate pain. This is highly problematic given that a number of chronic pain patients-those with interpersonal distress-often do not complete, and thus, do not benefit fully from existing treatments. Even if treatment is completed, individuals may not maintain improvements if they return to distressed social environments that undermine individual coping efforts. Thus, it is clear that new interventions derived from integrative models of individual and dyadic coping are needed to alleviate pain and suffering in patients who are at risk for poor treatment outcomes. This research study aims to develop a novel psychological intervention aimed at couples in which one partner has chronic pain. Our central hypothesis is that a theoretically integrative intervention that improves both partners' psychological flexibility (i.e., acceptance, mindfulness, values-based action) and relational flexibility (i.e., emotional disclosure, empathic responding) skills will be feasible and valid and that it will alleviate pain and improve quality of life. This is a departure from current practice, which focuses solely on the patient's individual functioning, does not address the spouse's psychological inflexibility, and does not address relationship issues.

ELIGIBILITY:
Inclusion Criteria:

* At least one spouse with some pain interference.
* Relationship dissatisfaction.
* Both partners at least 21 years old.
* Couples must also be married or cohabitating for at least 2 years regardless of sexual orientation to participate in the study.

Exclusion Criteria:

* Current suicidal or homicidal ideation or intent
* Current psychotic symptoms
* Cognitive impairment
* Malignancies (e.g., cancer) in either partner
* Current domestic violence

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-12; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in Depressive Symptoms from Baseline to 1-month Followup | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Beck Depression Inventory-II
Change in Pain Intensity | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Visual Rating Scale, Multidimensional Pain Inventory, Brief Pain Inventory
Change in Pain Quality | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  McGill Pain Questionnaire
Change in Quality of Life | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Satisfaction with Life Scale
Change in Relationship Satisfaction | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Dyadic Adjustment Scale; Dyadic Adjustment Scale-7
Change in Sleep Quality | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  PROMIS Sleep Disturbance and Sleep-related Impairment Scales
Change in Perceived Improvement | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Patient Global Impression of Change

SECONDARY OUTCOMES:
Change in Acceptance of Chronic Pain | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Chronic Pain Acceptance Questionnaire (baseline, post-treatment, followup); Chronic Pain Acceptance Chronic Pain Acceptance Questionnaire
Change in Anxiety and Catastrophizing about Pain | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Pain Anxiety Symptoms Scale, Pain Catastrophizing Scale (baseline, post-treatment, followup); Pain Catastrophizing Scale-Shortened Version (weekly)
Change in Mindfulness | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Five Facet Mindfulness Scale
Change in Values-Based Action | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Chronic Pain Values Inventory
Change in Dispositional Empathy | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Interpersonal Reactivity Index
Change in Emotional Expression | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Ambivalence Over Emotional Expression Questionnaire, Holding Back Scale
Change in Emotional Validation and Invalidation | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Coded from Couple Discussion Task
Change in Partner-perceived Empathy | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Perceived Partner Responsiveness Scale

OTHER OUTCOMES:
Treatment Credibility | Baseline
  Credibility of Treatment Scale
Therapist Adherence | Participants will be followed for the duration of the intervention, an expected average of 6 weeks
  audio recordings of sessions
Therapy Homework Compliance | Participants will be followed for the duration of the intervention, an expected average of 6 weeks
  Homework Rating Scale and time spend completing homework
Therapy Session Satisfaction | Participants will be followed for the duration of the intervention, an expected average of 6 weeks
  Participants' satisfaction with session
Intent to Complete Therapy Homework | Participants will be followed for the duration of the intervention, an expected average of 6 weeks
  Participants' intention to complete homework
Adverse Events | Participants will be followed for the duration of the intervention and followup period, an expected average of 10 weeks
  Adverse event data will be collected and reported

CONTACTS AND LOCATIONS:
Overall Officials: Annmarie Cano, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States